CLINICAL TRIAL: NCT03504930
Title: COLISURG Prospective, Multicentric Cohort of Ulcerative Colitis Requiring Surgical Treatment With Ileal Pouch-anal Anastomosis. Impact of Biotherapies on Sexual Function and Postoperative Morbidity.
Brief Title: COLISURG : Exploratory Analysis of Sexual Function and the Impact of Biotherapies on Postoperative Morbidity.
Acronym: COLISURG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0178
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
Keywords: Surgical; Ileal pouch-anal anastomosis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impact of biotherapy on postoperative morbidity: Impact of biotherapy on postoperative morbidity in ulcerative colitis
  Interventions: Other: Impact of biotherapy on postoperative morbidity in ulcerative colitis

INTERVENTIONS:
Other: Impact of biotherapy on postoperative morbidity in ulcerative colitis — Impact of biotherapy on postoperative morbidity, quality of life, sexual function, sexual health in ulcerative colitis

SUMMARY:
The surgical treatment of the ulcerative colitis (UC) remains associate to a significant morbidity (up to 60%). Anastomotic fistula and pelvic sepsis are the most severe complications which could dramatically compromise the surgical issue and functional status. Thanks to the current therapeutic arsenal and the evolution of health care paradigms, the quality of life of patients plays a key role in the modern global management of these medical conditions. Biotherapies (e.g anti-TNF) are widely used to treat patients with UC. Anti-TNF and anti-integrins have an effect on the immune response and can theoretically aggravate the infectious disease. Their potential impact on postoperative complications after ileo anal anastomosis (AIA) remains debated. Very few studies have looked at other biotherapies including vedolizumab. All studies are retrospective series with small sample size. Here again the conclusion remain contradictory. Lightner et al. showed an increased risk of surgical site infection for patients preoperatively exposed to vedolizumab (37% vs. 10%, p <0.001). In a dedicated cohort to the RCH, the same author found a risk of increased pelvic abscess (31.3% vs 5.9%, NS) but the difference was not statistically significant probably for lack of power. Other studies did not find any impact of vedolizumab on the risk of postoperative complications. To clearly determine within a large prospective cohort the impact of anti-TNF agents and biotherapies on the postoperative complications seems to be essential in order to adapt and to optimize the therapeutic strategy, especially the surgical sequences, in patients with UCR whom benefit a surgery.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 13 ans

- Patients with ulcerative colitis requiring surgical treatment with ileal pouch-anal anastomosis

Exclusion Criteria:

* Age < 13 ans
* Under any administrative or legal supervision

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ulcerative colitis requiring surgical treatment with ileal pouch-anal anastomosis
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Infectious complications at D30 postoperative | First month (Day 30) after surgery (Day 0)
  Infectious complications during the first month (D30) after surgery (D0)

CONTACTS AND LOCATIONS:
Overall Officials: Eddy COTTE, MD, Principal Investigator — Hospices Civils de Lyon; Quentin DENOST, MD, Principal Investigator — University Hospital, Bordeaux
Locations (22):
- France (22):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - APHP - Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Lille, Lille
  - APHM - Hôpital Nord, Marseille
  - Centre Hospitalier Universitaire de Nice - Hôpital L'Archet II, Nice
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital Européen Georges Pompidou, Paris
  - APHP - Hôpital St Antoine, Paris
  - APHP - Hôpital St Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon SUD, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier Universitaire de Tours, Tours
  - Centre Hospitalier Universitaire de Nancy, Vandœuvre-lès-Nancy